CLINICAL TRIAL: NCT02835092
Title: A Randomized, Controlled, 3-Arm Clinical Trial to Assess Weight Loss Using the Take Shape For Life Program or the Medifast Direct Program Versus a Self-Directed Diet
Brief Title: Weight Loss Using the Take Shape For Life Program or the Medifast Direct Program Versus a Self-Directed Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medifast, Inc. (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-1607 (MED 019)
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Self-directed Control (Active Comparator)
  Interventions: Other: Self-directed Control
- Take Shape For Life Program (Experimental)
  Interventions: Other: Take Shape For Life Program
- Medifast Direct Program (Experimental)
  Interventions: Other: Medifast Direct Program

INTERVENTIONS:
Other: Take Shape For Life Program — The Take Shape For Life (TSFL) Program group will be assigned to the Optimal Weight 5 & 1 Plan™ for weight loss. This group will have scheduled coaching sessions with a TSFL coach for the duration of the study.
  Arms: Take Shape For Life Program
Other: Medifast Direct Program — The Medifast Direct Program (MEDD) group will be assigned to the Medifast Achieve™ Plan (4 & 2 & 1 Plan®) for weight loss. MEDD participants will have access to the services of the Medifast Nutrition Support Team.
  Arms: Medifast Direct Program
Other: Self-directed Control — The Self-directed Control Group will be assigned to a food-based, reduced calorie diet consistent with the 2015 Dietary Guidelines for Americans.
  Arms: Self-directed Control

SUMMARY:
The study evaluates the effects of two commercially available weight loss programs, the TSFL and the MEDD programs, each compared to a self-directed control diet, on changes in body weight over a 16-week weight loss phase, in apparently healthy overweight and obese men and women.

ELIGIBILITY:
Inclusion Criteria:

* Participant is judged by the Clinical Investigator to be in good health on the basis of medical history and screening laboratory assessments.
* Participant has a BMI of 27.0 to 42.0 kg/m2 at start of intervention.
* Participant has no plans to change smoking habits during the study period.
* Participant is willing and able to comply with the visit schedule.
* Participant is willing to modify their physical activity level in accordance with recommendations provided with each group.
* In the Clinical Investigator's opinion, participant has interest in losing weight, and is ready and willing to do so.
* Participant is willing/able to follow assigned plan and adhere to food and beverage consumption guidelines for the duration of the study period.
* Participant has access to the internet via a computer, tablet, and/or smart phone.
* Participant understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Clinical Investigators.

Exclusion Criteria:

* Participant has an abnormal laboratory test result of clinical significance at the screening visit, at the discretion of the Clinical Investigator.
* Participant has had a weight loss or gain >5% in the 6 months prior to the screening visit except in the case of post-partum weight loss.
* Participant has extreme dietary habits, including vegetarianism, in the judgment of the Clinical Investigator.
* Participant has used medications, products, supplements, and/or programs/diets intended to alter body weight within 6 months of the screening visit.
* Participant has used medications which are known to stimulate or suppress appetite, and/or alter body weight but which are taken for other indications, will be allowed as long as the dose has remained stable for the past 6 months.
* Participant has used thyroid hormones, except stable-dose replacement therapy for ≥2 months prior to the screening visit.
* Participant has used Coumadin® (warfarin), and/or medications that may influence lipids and/or blood pressure, except stable-dose medications for 1 month prior to the screening visit.
* Participant has used medications that may influence carbohydrate metabolism, including but not limited to hypoglycemic medications and systemic (intravenous, intramuscular, or oral) corticosteroids within 1 month of the screening visit.
* Participant has used lithium within 1 month of the screening visit.
* Participant has a history of any surgery or liposuction for weight reducing purposes.
* Participant has a history or presence of clinically important gout, cardiac, renal, hepatic, endocrine (type 1 diabetes mellitus or type 2 diabetes mellitus that requires medication), pulmonary, biliary, pancreatic, or neurologic disorders.
* Participant has a history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa or binge eating) diagnosed by a health professional.
* Participant has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at screening visit.
* Participant has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Participant has elective hospitalizations planned (e.g., elective cosmetic procedures) during the study period.
* Participant is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
* Participant has a recent history of (within 12 months of Visit 1; week -1) or strong potential for alcohol or substance abuse. Alcohol abuse defined as >14 drinks/week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Participant has a known allergy, sensitivity, or intolerance to the study foods or any ingredient(s) of the study diets (e.g., soy, gluten, wheat, lactose).
* Exposure to any non-registered drug product within 1 month prior to the screening visit.
* Participant has a condition the Clinical Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Cook, PhD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-directed Control | Take Shape For Life Program | Medifast Direct Program
Started | 66 | 65 | 67
Completed | 63 | 57 | 64
Not Completed | 3 | 8 | 3
Not completed — Withdrawal by Subject | 3 | 6 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-directed Control | Take Shape For Life Program | Medifast Direct Program | Total
Number analyzed (Participants) | 66 | 65 | 67 | 198
Age, Continuous [Mean (Full Range); unit: years] | 46.3 [23 to 64] | 45.2 [20 to 64] | 45.7 [19 to 65] | 45.7 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 54 | 160
  Male | 12 | 13 | 13 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 13 | 10 | 34
  White | 50 | 45 | 54 | 149
  More than one race | 2 | 3 | 0 | 5
  Unknown or Not Reported | 1 | 2 | 3 | 6
Weight [Mean (Full Range); unit: kg] | 93.90 [71.40 to 127.80] | 95.51 [69.30 to 135.30] | 95.80 [69.20 to 130.20] | 95.07 [69.20 to 135.30]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 33.81 [28.40 to 41.70] | 34.49 [28.10 to 43.30] | 34.20 [27.40 to 41.90] | 34.16 [27.40 to 43.30]

OUTCOME MEASURES:

1. Primary Outcome: Body Weight Change
Description: Body weight (in gown, without shoes) was measured at each clinic visit on a medical quality digital scale (Health-o-meter 349KLX, Pelstar, McCook, IL) following a 10-14-hr fast. The relevant time points to determine body weight change were baseline and 16 weeks. The value for body weight at 16 weeks minus the value at baseline was the calculation used to determine body weight change.
Time Frame: 16 weeks
Population: Intent-to-Treat population, includes all participants randomized into the study.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Self-directed Control | Take Shape For Life Program | Medifast Direct Program
Number analyzed (Participants) | 66 | 65 | 67
kg | -0.23 (0.39) | -5.13 (0.86) | -4.98 (0.69)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: All intervention-emergent adverse events (AEs) occurring after randomization were collected at each clinic visit for assessment of safety.
Arm/Group | Self-directed Control | Take Shape For Life Program | Medifast Direct Program
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/65 | 0/67
Serious Adverse Events (participants affected / at risk) | 1/66 | 2/65 | 1/67
Other Adverse Events (participants affected / at risk) | 15/66 | 9/65 | 12/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-directed Control (N=66) | Take Shape For Life Program (N=65) | Medifast Direct Program (N=67)
Vertigo and Neck Strain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Partial Knee Orthoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-directed Control (N=66) | Take Shape For Life Program (N=65) | Medifast Direct Program (N=67)
Upper Respiratory Tract Infections (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 9 (9) | 8 (8)
Decreased frequency of bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT02835092/SAP_000.pdf
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT02835092/Prot_001.pdf